CLINICAL TRIAL: NCT05812222
Title: The Effect of Early Skin-to-Skin Contact in Normal Births on Suction Sufficiency, Stress and Bilirubin Levels of Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Nursing123456
Record Dates: First submitted 2023-04-02; First posted 2023-04-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-03

CONDITIONS: Nurse's Role; Breastfeeding
Keywords: skin-to-skin contact; normal delivery; stress; breastfeeding; jaundice
MeSH Terms: conditions — Breast Feeding; Jaundice

STUDY DESIGN:
Intervention Model Description: Intervention group and control group, randomized controlled, experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (skin-to-skin contact group) (Experimental): Skin-to-skin contact: It is the laying of the newborn in the prone position on the mother's bare chest area with only a diaper on.
  The stress levels of newborns were determined using the "Neonatal Stress Scale" immediately after birth, under a radiant heater, 5 minutes after SSC administration, and during IM K vit injection while SSC was administered (4 different time periods).
  The suction sufficiency of newborns was evaluated by the investigator using the "LATCH Breastfeeding Assessment Tool", 5 minutes after the initiation of early SSC immediately after birth, within the first hour after birth in the maternity ward, and 24 hours after birth.
  Interventions: Behavioral: Skin-to-Skin contact.
- control group (No Intervention): The routine applications of the hospital were applied to the mothers and newborns in the control group.
  The stress level of newborns was determined immediately after birth, under a radiant heater, and during IM K vit injection (3 different time periods) using the "Neonatal Stress Scale".
  The suction sufficiency of newborns within the first hour after birth and 24 hours after birth was evaluated by the researcher using the "LATCH Breastfeeding Assessment Tool".

INTERVENTIONS:
Behavioral: Skin-to-Skin contact. — Skin to skin contact: It is the laying of the newborn in the prone position on the mother's bare chest with only a diaper on.
  Arms: intervention group (skin-to-skin contact group)

SUMMARY:
Breastfeeding is one of the most effective ways to ensure a baby's health and survival, and breast milk is the ideal food for babies. It is recommended to start breastfeeding within the first hour of life, following skin-to-skin contact between the mother and the newborn immediately after birth.

Newborns transition from the dark, narrow and fluid-filled intrauterine environment to the wide, bright, cold and dry extrauterine life during the birth process. Thus, in addition to invasive procedures such as heel lance, vascular access, etc., including the birth process, simple and routine procedures such as separation from its mother in a short time to measure body weight cause stress for the newborn. For this reason, it is recommended that newborns should not be separated from their mothers except for important medical reasons, and that skin-to-skin contact should be initiated as soon as possible after birth so that the newborn can cope with the "birth stress".

Hyperbilirubinemia, as physiological jaundice, usually begins in the first 24-72 hours of life in term newborns. It peaks in the following days and starts to decrease in the following days. Colostrum, which is a natural laxative found in breast milk, facilitates the removal of meconium in the newborn and provides bilirubin excretion with stool. With early skin-to-skin contact between mother and newborn in the first minutes of life after birth; Nurses have a key role in reducing the level of "birth stress" experienced by the newborn and in reducing the severity of hyperbilirubinemia by starting breastfeeding early.

DETAILED DESCRIPTION:
The aim of this study; The aim of this study is to examine the effect of early SSC applied after normal delivery on the newborn's sucking efficiency, postnatal stress and bilirubin levels.

Study hypotheses:

H1: Early skin-to-skin contact applied immediately after normal birth has an effect on the sucking efficiency of the newborn.

H2: Normal doğumdan hemen sonra uygulanan erken erken ten tene temasın yenidoğanın stres düzeyine etkisi vardır.

H3: Early skin-to-skin contact applied immediately after normal delivery has an effect on the newborn's bilirubin level.

Type of the research: The research was conducted in a randomized controlled experimental type. Mothers and newborns who met the inclusion criteria were randomly selected by tossing a coin and assigned to the intervention or control groups. The data were collected by the researcher by face-to-face interview method.

ELIGIBILITY:
Inclusion Criteria:

For mothers;

* Vaginal delivery planning,
* Be between the ages of 18-45,
* Having a singleton pregnancy
* Having completed the 37th week of gestation,
* Agreeing to participate in the research,
* Absence of breastfeeding barriers [without human T-cell lymphotropic virus (HTLV-1), human Immunodeficiency virus (HIV) and active tuberculosis]
* Absence of any known health problems (such as diabetes, gestational diabetes, hypertension, Preeclampsia, renal failure, cardiac problems, psychiatric disorders)
* There was no ABO and Rh incompatibility. For newborns;
* Absence of conditions that prevent sucking such as frenulum or palate problem,
* Absence of any health problems or congenital diseases,
* Apgar Score ≥ 8
* No need for resuscitation after birth.

Exclusion Criteria:

-

Ages: 2 Minutes to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
The effect of early skin-to-skin contact applied immediately after normal delivery on the sucking efficiency of the newborn. | through study completion, an average of 1 year
  "LATCH Breastfeeding Diagnostic Scale" was used to determine the effect of skin-to-skin contact on sucking efficiency of newborns.
  A high score from the scale shows that mothers have good breastfeeding success and newborns have good sucking success.
  The name of the "LATCH Breastfeeding Diagnostic Scale" consists of the English initials of the 5 assessment criteria; [L (Latch on the breast), A (Audible swallowing), T (Type of the nipple), C (Comfort breast/nipple), H (Hold)].
  The sucking efficiency of newborns was evaluated by the researcher with the "LATCH Breastfeeding Diagnostic Scale", 5 minutes after the initiation of early skin-to-skin contact immediately after birth, within the first hour after birth in the maternity ward, and 24 hours after birth.
The effect of early skin-to-skin contact applied immediately after normal delivery on the stress level of the newborn. | through study completion, an average of 1 year
  "Newborn Stress Scale" was used to determine the effect of skin-to-skin contact on after immediately normal delivery stress level of newborns.
  A minimum of 0 points and a maximum of 16 points are taken from the scale. As the score increases, the stress level of the newborn increases.
  The stress levels of newborns were determined using the "Neonatal Stress Scale" immediately after birth, under a radiant heater, 5 minutes after SSC administration, and during IM K vit injection while SSC was administered (4 different time periods).
The effect of early skin-to-skin contact applied immediately after normal delivery on the bilirubin level of the newborn. | through study completion, an average of 1 year
  Starting breastfeeding at least 5 minutes after the skin-to-skin contact application and feeding only with breast milk in the following days.
  The determination of feeding only breast milk and formula, body weight and total serum bilirubin level of a newborn brought to the hospital by her parents for routine control on the fifth day of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)